CLINICAL TRIAL: NCT04930224
Title: Comparing the Impact of Serum GPER-1 and Oxidant/Antioxidant Levels on Retinopathy in Diabetic Patients and Healthy Individuals: A Pilot Study
Brief Title: Serum GPER-1 and Oxidant/Antioxidant Levels on Retinopathy in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Abdullah Beyoğlu, Assist of Prof, Kahramanmaras Sutcu Imam University
Other Study IDs: (Project no: 2019/5-24 M
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Hormones
Keywords: Diabetic retinopathy; GPER-1; oestradiol; progesterone; TSH; oxidative stress; neuronal damage.
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Proliferative Diabetic retinopathy: 40 patients with proliferative diabetic retinopathy
  Interventions: Diagnostic Test: The effect of GPER-1 on the formation of diabetic retinopathy
- Non-Proliferative Diabetic retinopathy: 40 patients with non-proliferative diabetic retinopathy
  Interventions: Diagnostic Test: The effect of GPER-1 on the formation of diabetic retinopathy
- Healthy individuals: 40 healthy persons
  Interventions: Diagnostic Test: The effect of GPER-1 on the formation of diabetic retinopathy

INTERVENTIONS:
Diagnostic Test: The effect of GPER-1 on the formation of diabetic retinopathy — Demonstrating the neuroprotective effect of GPER-1 in the formation of diabetic retinopathy and being a guide for new treatment models

SUMMARY:
Observational, comparative, cross-sectional study

DETAILED DESCRIPTION:
This study was conducted on G protein-mediated estrogen receptor 1 (GPER-1), which is thought to be effective in preventing the development of diabetic retinopathy (DR). There are studies proving that GPER-1 prevents neuroprotective effects and vascular pathology in many tissues. In the study, serum GPER-1 and oxidative stress biomarker levels were compared in diabetic patients and healthy control groups. GPER-1 was found to be significantly increased in diabetic patients. In addition, a positive correlation was found with oxidant markers. This may lead to new treatment models in the future.

ELIGIBILITY:
Inclusion Criteria:

* 40 individuals were required to have Proliferative Diabetic Retinopathy (PDR);
* 40 were required to have Non-PDR;
* 40 were required to be healthy, without any systemic disease.

Exclusion Criteria:

* Glaucoma,
* Ocular trauma sequelae,
* Pathological myopia,
* Non-diabetic retinopathy,
* A history of previous ocular surgery,
* Endocrine disorders (e.g.,thyroidopathy, adrenal gland disorders, pituitary pathologies),
* Opacities interfering with fundus examination (e.g., corneal opacity, lens opacity, vitreous cloudiness other than diabetic haemorrhage).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who applied to the tertiary eye outpatient clinic
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
G receptor-mediated protein-1 (GPER-1) | Baseline
  Variation of GPER-1 during the development of diabetic retinopathy
Oxidative/antioxidative stress markers (malondialdehyde [MDA]) | Baseline
  Variation of oxidative/antioxidative stress markers during the development of diabetic retinopathy
Oxidative/antioxidative stress markers (catalase [CAT]) | Baseline
  Variation of oxidative/antioxidative stress markers during the development of diabetic retinopathy
Oxidative/antioxidative stress markers (superoxide dismutase [SOD] | Baseline
  Variation of oxidative/antioxidative stress markers during the development of diabetic retinopathy
Thyroid stimulating hormone (TSH) | Baseline
  Variation of TSH during the development of diabetic retinopathy
Progesterone | Baseline
  Variation of progeterone during the development of diabetic retinopathy
oestradiol | Baseline
  Variation of oestradiol during the development of diabetic retinopathy

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Beyoğlu, MD, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Abdullah Beyoğlu, Kahramanmaraş, None Selected, Turkey (Türkiye)